CLINICAL TRIAL: NCT01712880
Title: The Treatment of the Acute Periprosthetic Hip Infection After Uncemented Total Hip Arthroplasty: A Randomized Study Comparing Open Debridement Component Retention (ODCR) With Modular Exchange Versus One Stage Exchange Arthroplasty
Brief Title: Treatment of Acute Periprosthetic Total Hip Arthroplasty Infections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not feasible.
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Midwest Orthopaedics at Rush (Other); University of California, San Francisco (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12055
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Periprosthetic Infection Total Hip Arthoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open debridement with modular exchange (Active Comparator)
  Interventions: Procedure: open debridement with modular exchange
- one stage exchange (Active Comparator)
  Interventions: Procedure: one stage exchange

INTERVENTIONS:
Procedure: open debridement with modular exchange
  Arms: open debridement with modular exchange
Procedure: one stage exchange
  Arms: one stage exchange

SUMMARY:
The purpose of this study is to determine the success rate of two treatments for infection after total hip replacement: single stage arthroplasty exchange (your surgeon will take out your original implants and replace them with a complete new set) compared to irrigation and debridement with modular exchange (your surgeon will clean your implants with a surgical solution and take out the plastic liner and replace it with a new one - the rest of your hip implants will stay in place). The goal is to see if one is better than the other for the treatment of hip infection after a total hip replacement. A successful treatment means that you did not have to have another surgery on your hip for an infection-related reason.

ELIGIBILITY:
Inclusion Criteria:

1. Return to the OR for a drainage procedure within six weeks of index primary uncemented arthroplasty 1a) Exam findings within six weeks of index operation:

   * Drainage for more than 7 days
   * Wound appearance consistent with deep infection or hematoma
   * Persistent fever or evidence of bacteremia
   * All patients currently deemed appropriate for irrigation and debridement
2. Labs

   - Rising inflammatory seromarkers
3. Aspiration with a positive culture

Exclusion Criteria:

1. Previous history of periprosthetic infection
2. Prisoners
3. Patients not willing to consent for the proposed treatment
4. Patients with altered mental status
5. Concurrent metastatic infection
6. Superficial Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Success | 2 year
  Success is defined as no subsequent revision surgery needed to treat chronic or acute periprosthetic infection

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institue, Charlotte, North Carolina, United States